CLINICAL TRIAL: NCT05891353
Title: Pain Modulatory Profiles in Stretching in Healthy Participants
Brief Title: Pain Modulatory Profiles in Stretching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Abigail Wilson, Assistant Professor, University of Central Florida
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2023-05-22; First posted 2023-06-06 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cold Water Immersion (Active Comparator): Participants will complete a cold water immersion task to the hand for one minute, four times. Change in Pressure Pain Threshold will be measured between each one-minute interval on the web space of the foot between the first and second toes.
  Interventions: Other: Cold Water Immersion
- Pain Inducing Stretch (Experimental): Participants will be seated in a chair and asked to complete an upper trapezius stretch. They will feel a gentle stretch in the area between the top of their shoulder and the base of their neck. Participants will be asked to stretch until the point of pain. They will hold this stretch for 1 minute, 4 times. Change in Pressure Pain Threshold will be examined on the web space of their foot between each one minute interval of the stretch. Participants will be notified that they may stop the stretch at any point if needed.
  Interventions: Other: Pain Inducing Stretch
- Pain Free Stretch (Active Comparator): Participants will be seated in a chair and asked to complete an upper trapezius stretch. They will feel a gentle stretch in the area between the top of their shoulder and the base of their neck. Participants will be asked to stretch in a pain free range. They will hold this stretch for 1 minute, 4 times. Change in Pressure Pain Threshold will be examined on the web space of their foot between each one minute interval of the stretch. Participants will be notified that they may stop the stretch at any point if needed.
  Interventions: Other: Pain Free Stretch

INTERVENTIONS:
Other: Cold Water Immersion — Cold Water Immersion task of hand
  Arms: Cold Water Immersion
Other: Pain Inducing Stretch — Moderately painful stretch of the neck
  Arms: Pain Inducing Stretch
Other: Pain Free Stretch — Pain free stretch of the neck
  Arms: Pain Free Stretch

SUMMARY:
The purpose of this study is to characterize immediate changes in pain sensitivity during stretching to the point of pain, stretching in a pain free range, and a cold water immersion task. Participants will attend three sessions during which they will undergo pain sensitivity assessment and complete the assigned intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pain Free

Exclusion Criteria:

* Non-English speaking
* Regular use of prescription pain medications
* Current or history of chronic pain condition
* Currently taking blood-thinning medication
* Any blood clotting disorder, such as hemophilia
* Systemic medical condition known to affect sensation, such as uncontrolled diabetes or neurological conditions
* Any contraindication to the application of ice, such as: uncontrolled hypertension, cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, circulatory compromise
* Not physically ready to exercise without a medical exam as indicated by the Physical Activity Readiness Questionnaire Plus (PAR-Q+)
* Surgery, injury, or fracture to the neck or upper extremity within the past 6 months
* Unable to perform the stretch
* Unable to attend all three sessions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Cold Water Immersion, Pain Inducing Stretch, Pain Free Stretch: Participants will complete a cold water immersion task to the hand for one minute, four times. Change in Pressure Pain Threshold will be measured between each one-minute interval on the web space of the foot between the first and second toes.
  For the pain inducing stretch, participants will be seated in a chair and asked to complete an upper trapezius stretch. They will feel a gentle stretch in the area between the top of their shoulder and the base of their neck. Participants will be asked to stretch until the point of pain. They will hold this stretch for 1 minute, 4 times. Change in Pressure Pain Threshold will be examined on the web space of their foot between each one minute interval of the stretch. Participants will be notified that they may stop the stretch at any point if needed.
  For the pain free stretch, participants will be seated in a chair and asked to complete an upper trapezius stretch. They will feel a gentle stretch in the area between the top of their shoulder and the base of their neck. Participants will be asked to stretch in a pain free range. They will hold this stretch for 1 minute, 4 times. Change in Pressure Pain Threshold will be examined on the web space of their foot between each one minute interval of the stretch. Participants will be notified that they may stop the stretch at any point if needed.
Period: Overall Study
Arm/Group | Cold Water Immersion, Pain Inducing Stretch, Pain Free Stretch
Started | 30
Completed Cold Water Immersion | 30
Completed Pain Inducing Stretch | 29
Completed Pain Free Stretch | 30
Completed | 29
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Cold Water Immersion, Pain Inducing Stretch, Pain Free Stretch: Participants will complete a cold water immersion task to the hand for one minute, four times. Change in Pressure Pain Threshold will be measured between each one-minute interval on the web space of the foot between the first and second toes.
  Cold Water Immersion: Cold Water Immersion task of hand
  Participants will be seated in a chair and asked to complete an upper trapezius stretch. They will feel a gentle stretch in the area between the top of their shoulder and the base of their neck. Participants will be asked to stretch until the point of pain. They will hold this stretch for 1 minute, 4 times. Change in Pressure Pain Threshold will be examined on the web space of their foot between each one minute interval of the stretch. Participants will be notified that they may stop the stretch at any point if needed.
  Pain Inducing Stretch: Moderately painful stretch of the neck
  Participants will be seated in a chair and asked to complete an upper trapezius stretch. They will feel a gentle stretch in the area between the top of their shoulder and the base of their neck. Participants will be asked to stretch in a pain free range. They will hold this stretch for 1 minute, 4 times. Change in Pressure Pain Threshold will be examined on the web space of their foot between each one minute interval of the stretch. Participants will be notified that they may stop the stretch at any point if needed.
  Pain Free Stretch: Pain free stretch of the neck
Arm/Group | Cold Water Immersion, Pain Inducing Stretch, Pain Free Stretch
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.88 (4.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Pressure Pain Threshold
Description: A pressure algometer will be applied between the first and second toe until the pressure sensation first becomes painful. Pressure pain threshold is applied between each one minute interval of the intervention.
Time Frame: Change in PPT is applied between minutes 1 and 4
Measure: Mean (Standard Deviation); unit: kilopascals
Arm/Group | Cold Water Immersion, Pain Inducing Stretch, Pain Free Stretch
Number analyzed (Participants) | 30
kilopascals
  Cold Water Immersion | 317.27 (137.27)
  Pain Inducing Stretch | 286.73 (154.48)
  Pain Free Stretch | 304.69 (145.05)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Cold Water Immersion, Pain Inducing Stretch, Pain Free Stretch
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT05891353/Prot_SAP_000.pdf